CLINICAL TRIAL: NCT00927602
Title: The Safety and Efficacy of Fondaparinux 1,5 mg for the Prevention of Venous Thromboembolism in Medical Patients With Renal Insufficiency
Brief Title: Fondaparinux 1,5 mg for the Prevention of Venous Thromboembolism (VTE) in Medical Patients With Renal Insufficiency
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: study was stopped after enrolment of about 200 patients for slow recruitment
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Walter Ageno, Associate Professor of Internal Medicine, Università degli Studi dell'Insubria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2008-005234-79
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Medical Patients; Renal Insufficiency
Keywords: renal failure; medical patient; venous thromboembolism; prophylaxis; fondaparinux
MeSH Terms: conditions — Renal Insufficiency; Venous Thromboembolism | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fondaparinux (Experimental)
  Interventions: Drug: fondaparinux

INTERVENTIONS:
Drug: fondaparinux — once daily sc injection, 1,5 mg, max 14 days
  Other Names: Arixtra

SUMMARY:
Fondaparinux is a parenteral anticoagulant drug and is approved for the prevention of venous thromboembolism in high risk medical patients. A relevant proportion of medical patients have moderate to severe renal insufficiency, which is an independent risk factor for bleeding. This risk may be further increased when low molecular weight heparin or fondaparinux are administered in patients with severe renal insufficiency, defined by a creatinine clearance of lower than 30 mL/min. No clear indications are available to reduce such risk in patients who require thromboprophylaxis. A lower dose of fondaparinux, 1.5 mg daily, has been recently approved for the prevention of venous thromboembolism in the specific population of patients with a creatinine clearance between 20 and 50 mL/min (European Marketing Authorization). However, there are to our knowledge no clinical studies that have assessed the safety and efficacy of this reduced dosage in medical patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Acute medical disease requiring thromboprophylaxis according to international guidelines
* Anticipated immobilization of at least 4 days
* Renal insufficiency defined by creatinine clearance between 20 and 50 mL/min according the MDRD formula
* Written informed consent

Exclusion Criteria:

* Active bleeding or bleeding in the previous 3 months
* Known bleeding diathesis
* Platelet count < 100.000
* Ongoing treatment with unfractionated heparin, low molecular weight heparin, fondaparinux, or vitamin K antagonists
* Use of prophylactic doses of heparin, low molecular weight heparin, or fondaparinux in the previous 72 hours
* Life expectancy < 1 month

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
major bleeding | up to 48 hours from last injection

SECONDARY OUTCOMES:
symptomatic venous thromboembolism | last treatment dose

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ageno, MD, Study Chair — Università degli Studi dell'Insubria; Francesco Dentali, MD, Study Director — Università degli Studi dell'Insubria; Alessandro Squizzato, MD, Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- University Of Insubria, Varese, Italy

REFERENCES:
- [Background] Cohen AT, Davidson BL, Gallus AS, Lassen MR, Prins MH, Tomkowski W, Turpie AG, Egberts JF, Lensing AW; ARTEMIS Investigators. Efficacy and safety of fondaparinux for the prevention of venous thromboembolism in older acute medical patients: randomised placebo controlled trial. BMJ. 2006 Feb 11;332(7537):325-9. doi: 10.1136/bmj.38733.466748.7C. Epub 2006 Jan 26. PMID 16439370
- [Background] Lim W, Dentali F, Eikelboom JW, Crowther MA. Meta-analysis: low-molecular-weight heparin and bleeding in patients with severe renal insufficiency. Ann Intern Med. 2006 May 2;144(9):673-84. doi: 10.7326/0003-4819-144-9-200605020-00011. PMID 16670137
- [Derived] Ageno W, Riva N, Noris P, Di Nisio M, La Regina M, Arioli D, Ria L, Monzani V, Cuppini S, Lupia E, Giorgi Pierfranceschi M, Dentali F; FONDAIR study group. Safety and efficacy of low-dose fondaparinux (1.5 mg) for the prevention of venous thromboembolism in acutely ill medical patients with renal impairment: the FONDAIR study. J Thromb Haemost. 2012 Nov;10(11):2291-7. doi: 10.1111/j.1538-7836.2012.04908.x. PMID 22925036